CLINICAL TRIAL: NCT06125340
Title: Optimizing Care for Children Hospitalized With Community-acquired Pneumonia: a Feasibility Randomized Controlled Trial of Short-course Antibiotic Therapy
Brief Title: Optimizing Care for Children Hospitalized With Community-acquired Pneumonia: Short-course Therapy
Acronym: PRESTO-2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jeffrey (Other)
Responsible Party: Sponsor-Investigator, Jeffrey, Associate Professor, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HHS-CB 2023-Pernica-2
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-04

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants in all arms will receive 5 days of study medications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short-course treatment (Experimental): 5 days of placebo (after participants already received 3-5 days of antibiotics)
  Interventions: Drug: Placebo
- Standard-duration treatment (Active Comparator): 5 days of amoxicillin (after participants already received 3-5 days of antibiotics)
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Placebo — 5 days of placebo to be given after 3-5 days of antibiotics
  Arms: Short-course treatment
Drug: Amoxicillin — Standard-dose amoxicillin (approved by Health Canada) to be given x 5 days.
  Arms: Standard-duration treatment

SUMMARY:
Children are commonly hospitalized because of community-acquired pneumonia (CAP). There are multiple high-quality randomized trials of short-course antibiotic therapy (3-5 days of treatment) for adults hospitalized with CAP - but there is very little evidence in children. We intend to do a pilot RCT of short-course (3-5 days) vs standard-duration (8-10 days) antibiotic therapy for children hospitalized for CAP.

ELIGIBILITY:
Inclusion Criteria:

* - children with a history of fever who are hospitalized with CAP (ie. 'severe CAP') as per the clinical team and who have abnormal chest imaging (eg. radiograph, ultrasound) will be eligible. They must also have at least one of the following:

  1. documented tachypnoea (>60 bpm for age <1 y, >50 bpm for 1-2 y, >40 bpm for 2-4 y, and >30 bpm for >4 y);
  2. cough on exam or by history;
  3. increased work of breathing on exam; or
  4. auscultatory findings (eg. focal crackles, bronchial breathing) consistent with CAP.

Exclusion Criteria:

* Children will be excluded if: antibiotics have been discontinued; they received >3 days of effective antibiotic treatment (excluding macrolide treatment) prior to hospitalization; there is supplemental oxygen use or fever within the past 24 h; more than 5 days elapsed since admission; the attending clinical team does not wish to use oral amoxicillin for treatment (because of allergy or any other reason); or the child is taking coumadin-based anticoagulants or tetracycline-type antibiotics (because of potential interactions with amoxicillin). Children will also be excluded if they have any of the following: chronic lung disease, congenital heart disease (requiring treatment or with exercise restrictions), malignancy, immunodeficiency (primary, acquired, or iatrogenic), a separate episode of pneumonia previously diagnosed within the past 2 weeks, or lung abscess diagnosed within the past six months. Children will not be eligible to participate more than once.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Consent success | Day 0
  The proportion of potentially eligible participants who consent
Open-label antibiotic use | before Day 30
  The proportion of participants who receive open-label (non-study) antibiotics
Losses to followup | before Day 30
  The proportion of participants lost to follow-up

SECONDARY OUTCOMES:
Proportion of participants with late clinical response | Day 15
  LCR is defined as:
  i) clinical improvement in fever, work of breathing, oral intake, and activity level, AND ii) lack of receipt of additional antimicrobials
Proportion of participants with repeat hospitalization for CAP | before Day 30
Proportion of participants with drug-related AEs (any severity) | before Day 30
Proportion of participants with serious drug AEs | before Day 30
Proportion of participants with unscheduled ED or urgent care visits | before Day 30
Proportion of participants with unscheduled primary care visits | before Day 30
Proportion of participants who develop complicated pneumonia | before Day 30
  Complicated defined by effusion, empyaema, necrotizing pneumonia

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada